CLINICAL TRIAL: NCT00745459
Title: Phase III General Clinical Study of NPO-11 in Patients Undergoing Gastric Endoscopy (Open-label Study)
Brief Title: Phase III General Clinical Study of NPO-11 in Patients Undergoing Gastric Endoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Nihon Pharmaceutical Co., Ltd (Industry)
Responsible Party: Yasumasa Ogawa, Nihon Pharmaceutical Co., Ltd
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPO-11-01/S-01
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2010-11-09 (Estimated); Status verified 2010-11

CONDITIONS: Stomach Diseases
Keywords: Patients; undergoing; gastric; endoscopy
MeSH Terms: conditions — Stomach Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- N (Experimental): 20 mL NPO-11
  Interventions: Drug: NPO-11

INTERVENTIONS:
Drug: NPO-11 — 20 mL NPO-11

SUMMARY:
Patients who require gastric endoscopy, including the patient population* excluded from the phase III controlled clinical study of NPO-11, will receive an intragastric single dose of NPO-11 20 mL. The efficacy of NPO-11 as a premedication for endoscopy will be evaluated based on the percentage of patients having no gastric peristalsis at both 2 minutes post-dose and the end of endoscopy (primary outcome measure).

The safety of NPO-11 will be evaluated based on adverse events and adverse drug reactions (ADRs) observed between administration and seven days after administration.

Patient population excluded from the phase III controlled clinical study of NPO-11

* Patients with reflux esophagitis
* Patients with active gastric or duodenal ulcers
* Patients who undergo endoscopy under sedation
* Patients who undergo endoscopy with a scope of <9 mm in diameter

ELIGIBILITY:
Inclusion Criteria:

Inpatients or outpatients of either sex who meet criteria (1) and (2) below will be enrolled in the study. Patients have to provide written informed consent for voluntary participation in the study.

1. Patients who require gastric endoscopy (except for emergency endoscopy or endoscopy for comprehensive medical examination)
2. Patients who are older than 20 years at the time of consent

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from the study. The criteria (2) and (3) will be confirmed during endoscopy. Patients who meet any of these criteria will be withdrawn from the study at the time of confirmation.

1. Patients with a history of surgery to the stomach
2. Patients with severe gastric stenosis or deformation which makes observation of gastric peristalsis difficult
3. Patients with upper gastrointestinal bleeding which requires hemostasis
4. Patients on cancer treatment (chemotherapy or radiotherapy)
5. Patients with a history of shock or hypersensitivity to l-menthol or peppermint oil (mint oil)
6. Patients with a history of shock or hypersensitivity to lidocaine hydrochloride
7. Pregnant or lactating women, women of childbearing potential, or women who plan to become pregnant during the study
8. Patients who have been exposed to NPO-11
9. Patients who have received other investigational drugs within four months before consent or who are participating in other clinical studies
10. Patients otherwise ineligible for participation in the study in the investigator's or subinvestigator's opinion

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Presence or absence of gastric peristalsis (central evaluation by independent evaluator) No gastric peristalsis is defined as when patients have no gastric peristalsis at both 2 minutes post-dose and the end of endoscopy. | each evaluation point

SECONDARY OUTCOMES:
Change in gastric peristalsis (central evaluation by independent evaluator) Difficulty level of intragastric observation (evaluation by investigator) Adverse events and ADRs observed between administration and 7 ± 3 days after administration | each evaluation point

CONTACTS AND LOCATIONS:
Locations (4):
- Japan (4):
  - Chūbu
  - Kansai
  - Kanto
  - Shikoku